CLINICAL TRIAL: NCT03323450
Title: Cognitive Remediation Therapy for Brain Tumor Patients: Improving Working Memory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-17-13581
Record Dates: First submitted 2017-10-11; First posted 2017-10-27 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Glioma; Brain Tumor, Primary
Keywords: High grade gliomas (WHO grade III or IV); Low grade gliomas (WHO Grade II)
MeSH Terms: conditions — Glioma; Brain Neoplasms; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High grade gliomas(WHO grade III or IV; n=15) (Experimental): The two groups will follow identical study timelines. Participants will receive a 1 hour training session on CogMed® (PI or trained graduate student). Participants will complete 5 weeks of CogMed® training within their own home. It consists of 25 training sessions. Each session lasts 30-45 minutes.The study team will check in with participants once a week via phone or email. Brief neuropsychological evaluations will be conducted at 4 time points. Each assessment will take approximately 30-60 minutes. Each participant will receive a $25 gift card to the VCU medical center gift shop at two time points.
  Interventions: Behavioral: CogMed®
- Low grade gliomas(WHO grade II; n=15) (Experimental): The two groups will follow identical study timelines. Participants will receive a 1 hour training session on CogMed® (PI or trained graduate student). Participants will complete 5 weeks of CogMed® training within their own home. It consists of 25 training sessions. Each session lasts 30-45 minutes.The study team will check in with participants once a week via phone or email. Brief neuropsychological evaluations will be conducted at 4 time points. Each assessment will take approximately 30-60 minutes. Each participant will receive a $25 gift card to the VCU medical center gift shop at two time points.
  Interventions: Behavioral: CogMed®

INTERVENTIONS:
Behavioral: CogMed® — It consists of 25 training sessions which can all be completed online and at home. Each session lasts 30-45 minutes. They must have a computer at home compatible with the CogMed® program.
  Brief neuropsychological evaluations will be conducted at 4 time points (these assessments are standard of care):
  1. Baseline before the participant is introduced to the CogMed® training program
  2. Within 2 weeks of completion of the CogMed® program
  3. At 3 months of completion of the CogMed® program to establish maintenance of gains
  4. At 6 months of completion of the CogMed® program to establish longer-term maintenance of gains

SUMMARY:
To investigate a computer-based Cognitive Remediation Therapy (CRT) for brain tumor patients at the Massey Cancer Center on measures of cognitive functioning (e.g., working memory, attention, processing speed, language, visuospatial functioning, immediate and delayed memory, or executive functioning) over time.

DETAILED DESCRIPTION:
Participants will be recruited by their neuropsychologist in the VCU Massey Cancer Center following standard neuropsychological evaluation (their neuro-oncologist may refer them to this study). If meeting inclusion criteria (described in later sections on participants), participants will be recruited and enrolled in the study. Two groups will be formed: High grade gliomas (WHO grade III or IV; n=15) and Low grade gliomas (WHO grade II; n=15). Participants will be followed over 11 months. The two groups will follow identical study timelines.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed primary brain tumor diagnosis via MRI and their neuro-oncologist
* A minimum of 2 months post-surgical resection or biopsy(if applicable)
* and/or a minimum 1 month post radiation treatment (if applicable)
* Karnofsky performance status more than 60
* Estimated intelligence at least 80 (standard score)
* Demonstrated attention difficulties (T-score of at least 65 on attention questionnaire or 1 or more standard deviations below mean on direct attention measures)
* No history of cognitive disorder
* No history of mood disorder
* Predicted life expectancy of at least 12 months
* Computer capability at home or provided a departmental iPad Mini to borrow for study purposes
* Primarily English speaking
* Aged 18+ (for which there is available age-adjusted neuropsychological testing standardization / normative data)

Exclusion Criteria:

* If they are not patients of Massey Cancer Center or do not meet the inclusion criteria listed above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Treatment enrollment rates | 6 months
  Determine feasibility and acceptability of the CogMed training program by assessing treatment enrollment
Attrition rates | 6 months
  Determine feasibility and acceptability of the CogMed training program by assessing attrition rates.
Change in scores on Behavior Rating Inventory of Executive Function-Adult (BRIEF-A) over time | Baseline to 6 months
  Brief neuropsychological evaluations will be conducted at 4 time points (these assessments are standard of care). Baseline before the participant is introduced to the CogMed® training program, within 2 weeks of completion of the CogMed® program, at 3 months of completion of the CogMed® program to establish maintenance of gains, and at 6 months of completion of the CogMed® program to establish longer-term maintenance of gains. During these time points, the scores are measured on Behavior Rating Inventory of Executive Function-Adult (BRIEF-A).
Change in scores on Conners' Continuous Performance Test - Third Edition (CPT-3) over time | Baseline to 6 months
  Brief neuropsychological evaluations will be conducted at 4 time points (these assessments are standard of care). Baseline before the participant is introduced to the CogMed® training program, within 2 weeks of completion of the CogMed® program, at 3 months of completion of the CogMed® program to establish maintenance of gains, and at 6 months of completion of the CogMed® program to establish longer-term maintenance of gains. During these time points, the scores are measured on Conners' Continuous Performance Test - Third Edition (CPT-3).
Change in scores on Delis-Kaplan Executive Function System (D-KEFS) over time | Baseline to 6 months
  Brief neuropsychological evaluations will be conducted at 4 time points (these assessments are standard of care). Baseline before the participant is introduced to the CogMed® training program, within 2 weeks of completion of the CogMed® program, at 3 months of completion of the CogMed® program to establish maintenance of gains, and at 6 months of completion of the CogMed® program to establish longer-term maintenance of gains. During these time points, the scores are measured on Delis-Kaplan Executive Function System (D-KEFS).
Change in scores on Repeatable Battery for the Assessment of Neuropsychological Status (RBANS-Update A, B, C, or D) over time | Baseline to 6 months
  Brief neuropsychological evaluations will be conducted at 4 time points (these assessments are standard of care). Baseline before the participant is introduced to the CogMed® training program, within 2 weeks of completion of the CogMed® program, at 3 months of completion of the CogMed® program to establish maintenance of gains, and at 6 months of completion of the CogMed® program to establish longer-term maintenance of gains. During these time points, the scores are measured on Repeatable Battery for the Assessment of Neuropsychological Status (RBANS-Update A, B, C, or D).
Scores on Test of Premorbid Functioning (TOPF) at baseline | Baseline
  Brief neuropsychological evaluations will be conducted at baseline before the participant is introduced to the CogMed® training program. During this time point, the scores are measured and compared on Test of Premorbid Functioning (TOPF) with other psychological measures.
Change in scores on Trial Making Test (TMT) over time | Baseline to 6 months
  Brief neuropsychological evaluations will be conducted at 4 time points (these assessments are standard of care). Baseline before the participant is introduced to the CogMed® training program, within 2 weeks of completion of the CogMed® program, at 3 months of completion of the CogMed® program to establish maintenance of gains, and at 6 months of completion of the CogMed® program to establish longer-term maintenance of gains. During these time points, the scores are measured on Trial Making Test (TMT).
Change in scores on Wechsler Memory Scale - Fourth Edition (WMS-IV) over time | Baseline to 6 months
  Brief neuropsychological evaluations will be conducted at 4 time points (these assessments are standard of care). Baseline before the participant is introduced to the CogMed® training program, within 2 weeks of completion of the CogMed® program, at 3 months of completion of the CogMed® program to establish maintenance of gains, and at 6 months of completion of the CogMed® program to establish longer-term maintenance of gains. During these time points, the scores are measured on Wechsler Memory Scale - Fourth Edition (WMS-IV).

SECONDARY OUTCOMES:
Change in scores on Beck Anxiety Inventory (BAI) over time | Baseline to 6 months
  Brief neuropsychological evaluations will be conducted at 4 time points (these assessments are standard of care). Baseline before the participant is introduced to the CogMed® training program, within 2 weeks of completion of the CogMed® program, at 3 months of completion of the CogMed® program to establish maintenance of gains, and at 6 months of completion of the CogMed® program to establish longer-term maintenance of gains. During these time points, the scores are measured on Beck Anxiety Inventory (BAI).
Change in scores on Beck Depression Inventory-II (BDI-II) over time | Baseline to 6 months
  Brief neuropsychological evaluations will be conducted at 4 time points (these assessments are standard of care). Baseline before the participant is introduced to the CogMed® training program, within 2 weeks of completion of the CogMed® program, at 3 months of completion of the CogMed® program to establish maintenance of gains, and at 6 months of completion of the CogMed® program to establish longer-term maintenance of gains. During these time points, the scores are measured on Beck Depression Inventory-II (BDI-II).

CONTACTS AND LOCATIONS:
Overall Officials: Ashlee Loughan, PhD, Principal Investigator — Massey Cancer Center
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States

REFERENCES:
- [Derived] Braun SE, Aslanzadeh FJ, Lanoye A, Fountain-Zaragoza S, Malkin MG, Loughan AR. Working memory training for adult glioma patients: a proof-of-concept study. J Neurooncol. 2021 Oct;155(1):25-34. doi: 10.1007/s11060-021-03839-y. Epub 2021 Sep 7. PMID 34491526